CLINICAL TRIAL: NCT02455817
Title: REWARDS-Angina at Follow up Post Stenting
Status: Withdrawn | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REWARDS- Angina
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2018-06

CONDITIONS: Rate of Angina

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Cypher: Access rate of angina including degree, post PCI up to 1 year for the Cypher stent.
- Taxus Express: Access rate of angina including degree, post PCI up to 1 year for the Taxus Express stent.
- Xience V: Access rate of angina including degree, post PCI up to 1 year for the Xience V stent.
- Promus Element: Access rate of angina including degree, post PCI up to 1 year for the Promus stent.
- Resolute: Access rate of angina including degree, post PCI up to 1 year for the Resolute stent.
- Bare metal stents: Access rate of angina including degree, post PCI up to 1 year for bare metal stents.

SUMMARY:
Single center, retrospective registry to collect data regarding the rate of angina (any and CCS clas III/IV) within 12 months post stent implantation. In addition, the target vessel revascularization rate within 12 months post stent implantation.

DETAILED DESCRIPTION:
The objective of this study is to retrospectively identify the rate of angina (any as well as CCS class III/IV) up to one (1) year following stent implantation. The following drug eluting stents will be evaluated in addition to bare metal stents; Cypher, Taxus Express, Xience V, Resolute and Promus Element. The target vessel revascularization rate will also be compared for the 6 stent types within one (1) year.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, > 18 years of age,
* Patients who received at least one (1) commercially available Drug Eluting Stent or Bare Metal Stent: Cypher, Taxus Express, Xience V, Promus Element, Resolute, or Bare Metal Stents

Exclusion Criteria:

* Received more than one type of DES as listed above or both a BMS and DES (as listed above)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients male or female, 18 years or older who have received at least one commercially available Drug Eluting Stent or Bare Metal Stent: Cypher, Taxus Express, Xience V, Promus Element, Resolute, or Bare Metal Stents
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Angina | up to 1 year
  post PCI for a variety of DES and BMS